CLINICAL TRIAL: NCT06496438
Title: Psychobiotics Ameliorate Anxiety and Depression Status in Patients Under Chemotherapy for Gastrointestinal Malignancies
Brief Title: Probiotics for Depression in Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ProDeCa
Record Dates: First submitted 2024-04-30; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-05

CONDITIONS: Depression; Anxiety Disorder; Probiotics; Gastrointestinal Cancer; Quality of Life; Chemotherapy
Keywords: Randomized Clinical Trial; Gastrointestinal Cancer; Chemotherapy; Psychobiotics; Depression; Anxiety; Quality of life
MeSH Terms: conditions — Depression; Anxiety Disorders; Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychobiotics (Active Comparator): Patients operated on for gastrointestinal cancer and currently undergoing chemotherapy will be randomized to receive a probiotic regime "therapy" with four psychobiotics [one sachet twice daily for a month].
  Interventions: Dietary Supplement: Psychobiotics
- Placebo (Placebo Comparator): Patients operated on for gastrointestinal cancer and currently undergoing chemotherapy will be randomized to receive placebo sachets which will be identical to the probiotic regime.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Psychobiotics — Dietary Supplement: A four probiotic regime, containing Lactobacillus rhamnosus, Bifidobacterium animalis subsp. lactis, Bifidobacterium breve, and Bifidobacterium longum at a concentration of 1, 000,000,000 CFU.
  Arms: Psychobiotics
Other: Placebo — The placebo regime, containing powdered glucose polymer, will be identical in packaging, appearance, consistency, and solubility in drinking water, thus making it impossible to recognize which are placebo and which the therapeutic formulation. Both will be identically standardized by the same pharmaceutical company [Uni-Pharma, Greece].
  Arms: Placebo

SUMMARY:
Anxiety and depressive disorders are quite prevalent in the general population. In 2015, it was estimated that 3.6% of the world population (around 264 million individuals) live with depression and 4.4% (around 322 million) with anxiety, while in the recent years of the COVID-19 pandemic, the prevalence of these disorders has significantly increased.

According to the American Psychiatric Association, in 2013 depression was defined as a serious mental illness characterized by decreased mood lasting more than 15 days, a lack of interest, and (even) apathy to normal daily activities. Depression, particularly in its severe form - the major depressive disorder (MDD), is the second leading cause of disability and the most common emotional disorder.

Recent research data indicate that this psychiatric disorder, as also similar neuropsychological conditions (Parkinson's, autism, etc.) have, as their main substrate, a disturbance in the diversity of the gut microbiome. More specifically, it has been shown that there is a direct and bidirectional communication between gut and brain - the "gut-brain-axis". The gut, through its microbiome, communicates with the brain by means of neural, immunological, and metabolic pathways, either directly, through the vagus nerve or indirectly, either through the microbiome immunomodulation or the tryptophan pathway, or by the production of various neuroactive molecules.

The disturbance in the diversity of the gut microbiome, termed dysbiosis, involves changes in the composition and the number of bacteria genera; and is causatively related to depression via the gut-brain axis. The transmission of nerve impulses, both via the hypothalamic-pituitary-adrenal axis and via the vagus nerve is disrupted by dysbiosis, leading to anxiety and depression, or, conversely, stressful conditions, more particularly emotional stress, which triggers an imbalance in the hypothalamic-pituitary-adrenal axis, leading to systemic immune responses and intestinal dysbiosis. This imbalance can clinically manifest with alterations in digestive tract function, knowledge accepted since the beginning of the previous century.

Nowadays, there is considerable evidence that the gut microbiome represents a novel anti-depressant and the term "psychobiotics" has been used to describe those species of probiotic bacteria excreting mental health benefits.

Certain Bifidobacterium and Lactobacillus species have already demonstrated, both experimentally and in clinical studies, their capability to improve mood, reduce anxiety, and enhance cognitive function. On these grounds, it is reasonable to raise the hypothesis that, by restoring the diversity of the gut microbiome, and thus enhancing the population of these specific probiotic species - termed 'psychobiotics', due to their specified functions, - could at least lead to an improvement in neuro-psychological disorders through gut-brain-axis remodeling.

DETAILED DESCRIPTION:
Based on the assumption that 1. at least one third of digestive cancer patients operated on - and probably more, when surgery is followed by chemotherapy sessions - suffer from anxiety and depression, 2. psychobiotics can beneficially modify the gut microbiome, 3. psychobiotics can improve the mental health of patients suffering from depression, and 4. there is no other study on the use of psychobiotics in anxiety and/or depression symptoms in patients operated on for digestive tract malignancies and subjected to chemotherapy thereafter the present study was designed to investigate the ability of a probiotic formulation containing bacteria with known psychobiotic properties to change the depression and anxiety status of digestive cancer patients undergoing chemotherapy postoperatively.

This study will be a prospective, double-blind, randomized study against placebo in patients operated on for digestive cancer and undergoing chemotherapy. The study will be conducted in the 1st Surgical Department of the Aristotle University of Thessaloniki, at the AHEPA University Hospital of Thessaloniki, Greece, in collaboration with the Outpatient Surgical Oncology Unit. Permission has already been obtained from the Scientific Council of the AHEPA Hospital (Approval Number: 313/4.7.2023).

The oncologist involved in the study protocol will be responsible for randomization. She will inform the patients who meet the study entry criteria of the purpose of the study, and receiving their written consent after detailed information. Patients having signed the informed consent will then be assigned at random [in a 1:1 ratio] to receive placebo or probiotic regime treatment, according to a computer-based table [randomized.com]. The randomization will be blinded to the study statistician, as well as to the physicians in contact with patients for interviews to facilitate the collection of answers to the questionnaires. Sealed envelops will be used to ensure blinding. Only the study coordinator will be aware of the content, having no further involvement with the patients. Each patient, having signed the consent, will then receive a unique code-number, being a combination of the anatomical location of the tumor, the patient's serial number, a capital letter A or B - blindly indicating the treatment groups - and a small letter, [a,b,c] indicating the physician who contacts each patient.

After patient aggrees to be included in the study, the demographic data that will be obtained in relation to each patient are: gender; age; body weight (in kilograms) and height (in meters) to calculate BMI; reported weight loss in kilograms since the disease diagnosis; marital status; smoking habits (no smoking or number of cigarettes/day); alcohol consumption (type and volume); and the possible use of tranquilizers [mg of active substance]. Optionally, patients will give information as to their educational level (1st, 2nd, or 3rd grade), annual income (<10.000€, 10.001-30.000€, >30.001€/year); and health care insurance (public, private, both). From their medical records cancer type and anatomical localization; cancer stage (TNM classification); type of surgical intervention; and co-morbidity indices (Charlson Comorbidity Index) will be obtained. Additional information will be collated relating to the time lapse since diagnosis (in days); the time lapse from hospital discharge to starting chemotherapy (in days); and the time from starting chemotherapy to study entry (in days).

The probiotic regime under testing is a combination of 4 psychobiotics: Lactobacillus rhamnosus, Bifidobacterium animalis subsp. lactis, Bifidobacterium breve, and Bifidobacterium longum, at a dose of 1.000.000.000/CFU. These for psychobiotics are the main ingredients of the commercially available formula LactoLevure®, ProbioMood [UniPharma, Athens, Greece], which also contains saffron and magnesium. This formula is marketed for "people with an anxious lifestyle who often suffer from symptoms such as low mood or fatigue as a result of stress".

The placebo regime, containing powdered glucose polymer, will be identical in packaging, appearance, consistency, and solubility in drinking water, thus making it impossible to recognize which are placebo and which the therapeutic formulation. Both will be identically standardized by the same pharmaceutical company [Uni-Pharma, Greece].

Patients will be administered the "treatment" or the placebo daily - one sachet twice a day, two hours after breakfast, for 30 consecutive days. At the follow-up appointment after treatment termination, patients will be required to return any remaining sachets which they forgot to take [Patients will be telephoned to remind a day before appointment). Fifteen days after the start of treatment, there will be telephone contact (or a face-to-face contact if the new chemotherapy appointment coincides) for the purpose of a rough, out of the protocol assessment of the patient's condition by the same physician who conducted the initial interview; the purpose being to confirm that the patient is receiving the treatment and to un-officially obtain information on whether he/she is generally feeling better than previously.

Two follow up evaluations will be held 1 month and 3 months, after treatment begins.

Patients will be evaluated by means of standardized questionnaires - officially translated and validated in the Greek language - for the quantification of depression, emotional state, anxiety, quality of life, physical weakness and pain.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and <85
* Histologically confirmed diagnosis of digestive tract malignancy, the tumor having been surgically resected and the patient currently undergoing chemotherapy sessions
* Informed consent obtained to participate in the study

Exclusion Criteria:

* Not understanding the Greek language
* Dementia
* Pre-existing psychiatric disorders
* Already receiving probiotic supplements (apart from yoghurt)
* Participation in another clinical trial
* Consumption of less than the 90% of treatment sachets/doses (verified by the sachets returned)
* Those having received during hospitalization other probiotic formulations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Depression changes | at one and 3 months
  To evaluate the ability of psychobiotics to change patients' depression status at one and 3 months [if available] after patients' recruitment in the study, against placebo treatment. The evaluation of patients' depression status will be performed with the help of Beck Depression Inventory Questionnaire (BDI) and Hamilton Depression Rating Scale (HAM-D). The total score of these questionnaires defines depression severity. BDI total score ranges from 0 to 63 and HAM-D total score ranges from 0 to 50. Regarding BDI a total score <10 reflects "mild" depression, 10-18 "mild to moderate", 19-29 "moderate to severe", and 30-63 "severe" depression and regarding HAM-D a total of score 0-7: reflects normal condition, 8-18: moderate depression, 19-22: severe depression, and 23-50: very severe depression. The total mean score differences will be compared between the probiotic and the placebo group for both questionnaires.

SECONDARY OUTCOMES:
Anxiety changes 1 | at one and 3 months
  To assess the efficacy of psychobiotics against placebo treatment to change anxiety status at one and 3 months [if available]. Anxiety will be assessed with the help of General Anxiety Disorder 7 (GAD-7) self-administered questionnaire. The questionnaire consists of seven items for which there are four response options "not at all", "several days", "more than half the days", and "nearly every day" being scored as 0, 1, 2, and 3, respectively. The patients are kindly requested to choose the proper answer based on how often each symptom occurred during the last two weeks. Then, the total score of the questionnaire is calculated. Cut off points of 5, 10, and 15 represent mild, moderate, and severe levels of anxiety, respectively, while total scores greater than 10 indicates potentially clinical condition. The total mean score differences will be compared between the probiotic and the placebo group.
Anxiety changes 2 | at one and 3 months
  To assess the efficacy of psychobiotics against placebo treatment to change anxiety status at one and 3 months [if available]. Additionally the Perceived Stress Scale - 14 items (PSS-14) will be administered. PSS-14 is self-administered questionnaire which consists of 14 items; 7 negative and 7 positives. The positive domain assesses the ability to deal with perceived stressors, while the negative element evaluates the loss of control, and pessimistic emotions or reactions. Each of the 14 items has a possible answer rated on a 5-point Likert-scale ranging from 0 ("never") to 4 ("very often"). After, the patient answers the questionnaire, the total score is calculated.
Health related quality of life changes | at one and 3 months
  To assess the efficacy of psychobiotics against placebo treatment to change health-related quality of life at one and 3 months [if available]. The assessment of health-related quality of life will be performed with the help of Medical Outcomes Study SF-36-Item Short Form Health Survey (SF-36) v1.0 questionnaire (SF-36). It consists of 36 items divided in 8 concepts/categories. For each item, responses were coded, summed and transformed into a scale ranging from 0 to 100; the higher the score the better health related quality of life status. The mean score for each one of the 8 concepts were measured. The total mean score differences will be compared between the probiotic and the placebo group.
Physical weakness changes | at one and 3 months
  To assess the efficacy of psychobiotics against placebo treatment to change physical weakness at one and 3 months [if available]. The physical weakness will be assessed based on the Clinical Frailty Scale (CFS) which was introduced in the second clinical examination of the Canadian Study of Health and Aging (CSHA) as a way to summarize the overall level of fitness or frailty of an older adult after they had been evaluated by an experienced clinician. CFS is 9-point scale (very fit, fit, managing well, living with very mild frailty, living with mild frailty, living with moderate frailty, loving with severe frailty, living with very severe frailty, terminally ill). Each patient will be evaluated by a physician and will be included in one of the aforementioned categories based on her/his physical status. The percent of patients including in each category will be recorded and compared between the probiotic and the placebo group.
Pain fellness changes | at one and 3 months
  To assess the efficacy of psychobiotics against placebo treatment to change pain fellness at one and 3 months [if available]. The Short-Form McGill Pain Questionnaire (SF-MPQ) will be used for the evaluation of pain. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0=none, 1=mild, 2=moderate or 3=severe. The higher the pain score the greater the pain. In addition, SF-MPQ also includes the Present Pain Intensity (PPI) index ranging from 0 to 5 (The higher the pain score the greater the pain) and a visual analogue scale (VAS) 100mm in length. The bigger the distance between the beginning of VAS and the cross made by the patient, the greater the magnitude of the patient's pain. The score ranges between 0 (minimum) and 100 (maximum). The total mean score differences will be compared between the probiotic and the placebo group.
Emotion Regulation changes | at one and 3 months
  Emotion Regulation Questionnaire (ERQ) was introduced by Gross and John in 2003 and it aims to assess the specific emotion regulation strategies that a person follows in order either to change the emotional impact or to inhibit an ongoing expressive behavior.
  The ERQ consists of two domains; the "Cognitive Reappraisal" and the "Expressive Suppression". The first dimension of ERQ evaluates the regulatory process of emotional controlling by changing the way of thinking about a certain situation, while the second one examines the strategy of suppressing emotions by not expressing them. Cognitive reappraisal is directly corelated with positive indicators, while expressive suppression with negative outcomes and depressive symptomatology. ERQ totally consists of ten items. Each item is scored on a 7-point Likert-type scale ranging from 1 to 7 (1: strongly disagree, 4: neutral, 7: strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Kotzampassi, Dr., Study Director — Aristotle University of Thessaloniki, Greece
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grassi L, Caruso R, Riba MB, Lloyd-Williams M, Kissane D, Rodin G, McFarland D, Campos-Rodenas R, Zachariae R, Santini D, Ripamonti CI; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Anxiety and depression in adult cancer patients: ESMO Clinical Practice Guideline. ESMO Open. 2023 Apr;8(2):101155. doi: 10.1016/j.esmoop.2023.101155. Epub 2023 Mar 14. PMID 37087199
- [Background] Sonali S, Ray B, Ahmed Tousif H, Rathipriya AG, Sunanda T, Mahalakshmi AM, Rungratanawanich W, Essa MM, Qoronfleh MW, Chidambaram SB, Song BJ. Mechanistic Insights into the Link between Gut Dysbiosis and Major Depression: An Extensive Review. Cells. 2022 Apr 16;11(8):1362. doi: 10.3390/cells11081362. PMID 35456041
- [Background] Butler MI, Sandhu K, Cryan JF, Dinan TG. From isoniazid to psychobiotics: the gut microbiome as a new antidepressant target. Br J Hosp Med (Lond). 2019 Mar 2;80(3):139-145. doi: 10.12968/hmed.2019.80.3.139. PMID 30860919
- [Background] Misra S, Mohanty D. Psychobiotics: A new approach for treating mental illness? Crit Rev Food Sci Nutr. 2019;59(8):1230-1236. doi: 10.1080/10408398.2017.1399860. Epub 2017 Nov 30. PMID 29190117
- [Background] Chidambaram SB, Essa MM, Rathipriya AG, Bishir M, Ray B, Mahalakshmi AM, Tousif AH, Sakharkar MK, Kashyap RS, Friedland RP, Monaghan TM. Gut dysbiosis, defective autophagy and altered immune responses in neurodegenerative diseases: Tales of a vicious cycle. Pharmacol Ther. 2022 Mar;231:107988. doi: 10.1016/j.pharmthera.2021.107988. Epub 2021 Sep 16. PMID 34536490
- [Background] Kim JK, Han SK, Joo MK, Kim DH. Buspirone alleviates anxiety, depression, and colitis; and modulates gut microbiota in mice. Sci Rep. 2021 Mar 17;11(1):6094. doi: 10.1038/s41598-021-85681-w. PMID 33731795
- [Background] Zhou L, Foster JA. Psychobiotics and the gut-brain axis: in the pursuit of happiness. Neuropsychiatr Dis Treat. 2015 Mar 16;11:715-23. doi: 10.2147/NDT.S61997. eCollection 2015. PMID 25834446
- [Background] O'Mahony SM, Marchesi JR, Scully P, Codling C, Ceolho AM, Quigley EM, Cryan JF, Dinan TG. Early life stress alters behavior, immunity, and microbiota in rats: implications for irritable bowel syndrome and psychiatric illnesses. Biol Psychiatry. 2009 Feb 1;65(3):263-7. doi: 10.1016/j.biopsych.2008.06.026. Epub 2008 Aug 23. PMID 18723164
- [Background] Naseribafrouei A, Hestad K, Avershina E, Sekelja M, Linlokken A, Wilson R, Rudi K. Correlation between the human fecal microbiota and depression. Neurogastroenterol Motil. 2014 Aug;26(8):1155-62. doi: 10.1111/nmo.12378. Epub 2014 Jun 1. PMID 24888394
- [Background] Mohammadi AA, Jazayeri S, Khosravi-Darani K, Solati Z, Mohammadpour N, Asemi Z, Adab Z, Djalali M, Tehrani-Doost M, Hosseini M, Eghtesadi S. The effects of probiotics on mental health and hypothalamic-pituitary-adrenal axis: A randomized, double-blind, placebo-controlled trial in petrochemical workers. Nutr Neurosci. 2016 Nov;19(9):387-395. doi: 10.1179/1476830515Y.0000000023. Epub 2015 Apr 16. PMID 25879690
- [Background] Johnson D, Letchumanan V, Thum CC, Thurairajasingam S, Lee LH. A Microbial-Based Approach to Mental Health: The Potential of Probiotics in the Treatment of Depression. Nutrients. 2023 Mar 13;15(6):1382. doi: 10.3390/nu15061382. PMID 36986112
- [Background] Messaoudi M, Lalonde R, Violle N, Javelot H, Desor D, Nejdi A, Bisson JF, Rougeot C, Pichelin M, Cazaubiel M, Cazaubiel JM. Assessment of psychotropic-like properties of a probiotic formulation (Lactobacillus helveticus R0052 and Bifidobacterium longum R0175) in rats and human subjects. Br J Nutr. 2011 Mar;105(5):755-64. doi: 10.1017/S0007114510004319. Epub 2010 Oct 26. PMID 20974015
- [Background] Rades D, Al-Salool A, Yu NY, Bartscht T. Emotional Distress Prior to Chemoradiation for Rectal or Anal Cancer. In Vivo. 2023 May-Jun;37(3):1205-1210. doi: 10.21873/invivo.13197. PMID 37103088
- [Background] Harms J, Kunzmann B, Bredereke J, Harms L, Jungbluth T, Zimmermann T. Anxiety in patients with gastrointestinal cancer undergoing primary surgery. J Cancer Res Clin Oncol. 2023 Sep;149(11):8191-8200. doi: 10.1007/s00432-023-04759-2. Epub 2023 Apr 15. PMID 37060473
- [Background] Die Trill M. Psychological aspects of depression in cancer patients: an update. Ann Oncol. 2012 Sep;23 Suppl 10:x302-5. doi: 10.1093/annonc/mds350. No abstract available. PMID 22987981
- [Background] Redeker NS, Lev EL, Ruggiero J. Insomnia, fatigue, anxiety, depression, and quality of life of cancer patients undergoing chemotherapy. Sch Inq Nurs Pract. 2000 Winter;14(4):275-90; discussion 291-8. PMID 11372188
- [Background] Zimmerman M, Martinez JH, Young D, Chelminski I, Dalrymple K. Severity classification on the Hamilton Depression Rating Scale. J Affect Disord. 2013 Sep 5;150(2):384-8. doi: 10.1016/j.jad.2013.04.028. Epub 2013 Jun 4. PMID 23759278
- [Background] Krebber AM, Buffart LM, Kleijn G, Riepma IC, de Bree R, Leemans CR, Becker A, Brug J, van Straten A, Cuijpers P, Verdonck-de Leeuw IM. Prevalence of depression in cancer patients: a meta-analysis of diagnostic interviews and self-report instruments. Psychooncology. 2014 Feb;23(2):121-30. doi: 10.1002/pon.3409. Epub 2013 Sep 16. PMID 24105788
- [Background] Kotzampassi K, Stavrou G, Damoraki G, Georgitsi M, Basdanis G, Tsaousi G, Giamarellos-Bourboulis EJ. A Four-Probiotics Regimen Reduces Postoperative Complications After Colorectal Surgery: A Randomized, Double-Blind, Placebo-Controlled Study. World J Surg. 2015 Nov;39(11):2776-83. doi: 10.1007/s00268-015-3071-z. PMID 25894405